CLINICAL TRIAL: NCT00099632
Title: Maintaining Options for Mothers Study (MOMS): A Phase II Randomized Comparison of Three Antiretroviral Strategies Administered for 7 or 21 Days to Reduce the Emergence of Nevirapine Resistant HIV-1 Following a Single Intrapartum Dose of Nevirapine
Brief Title: Comparison of Three Anti-HIV Regimens to Prevent Nevirapine Resistance in Women Who Take Nevirapine During Pregnancy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5207; 10127 (Registry Identifier: DAIDS ES); ACTG A5207; MOMS
Record Dates: First submitted 2004-12-17; First posted 2004-12-20 (Estimated); Results first posted 2012-01-19 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2019-01

CONDITIONS: HIV Infections
Keywords: Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; lamivudine, zidovudine drug combination; Lopinavir; Nevirapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 7-day 3TC/ZDV (Experimental): SD NVP and 3TC/ZDV provided at onset of active labor, followed by 7 days of 3TC/ZDV.
  Interventions: Drug: Lamivudine/Zidovudine; Drug: single dose Nevirapine
- 21-day 3TC/ZDV (Experimental): SD NVP and 3TC/ZDV provided at onset of active labor, followed by 21 days of 3TC/ZDV.
  Interventions: Drug: Lamivudine/Zidovudine; Drug: single dose Nevirapine
- 7-day FTC/TDF (Experimental): SD NVP and FTC/TDF provided at onset of active labor, followed by 7 days of FTC/TDF.
  Interventions: Drug: Emtricitabine/Tenofovir Disoproxil Fumarate; Drug: single dose Nevirapine
- 21-day FTC/TDF (Experimental): SD NVP and FTC/TDF provided at onset of active labor, followed by 21 days of FTC/TDF.
  Interventions: Drug: Emtricitabine/Tenofovir Disoproxil Fumarate; Drug: single dose Nevirapine
- 7-day LPV/r (Experimental): SD NVP and LPV/r provided at onset of active labor, followed by 7 days of LPV/r.
  Interventions: Drug: Lopinavir/Ritonavir; Drug: single dose Nevirapine
- 21-day LPV/r (Experimental): SD NVP and LPV/r provided at onset of active labor, followed by 7 days of LPV/r
  Interventions: Drug: Lopinavir/Ritonavir; Drug: single dose Nevirapine

INTERVENTIONS:
Drug: Emtricitabine/Tenofovir Disoproxil Fumarate — 200mg/300mg as one tablet taken orally once daily
  Other Names: FTC/TDF
  Arms: 21-day FTC/TDF; 7-day FTC/TDF
Drug: Lamivudine/Zidovudine — 150mg/300mg as one tablet taken orally twice daily
  Other Names: 3TC/ZDV
  Arms: 21-day 3TC/ZDV; 7-day 3TC/ZDV
Drug: Lopinavir/Ritonavir — 133.3mg/33.3mg as three capsules taken orally twice daily
  Other Names: LPV/r
  Arms: 21-day LPV/r; 7-day LPV/r
Drug: single dose Nevirapine — one 200 mg tablet taken orally
  Other Names: SD NVP

SUMMARY:
HIV infected pregnant women may take single-dose nevirapine (SD NVP) prior to giving birth to prevent mother-to-child transmission (MTCT) of HIV. However, SD NVP may cause NVP resistance in the mother, potentially ruling out some treatment options in the future. The purpose of this study is to determine which of three anti-HIV drug regimens most effectively reduces the development of maternal NVP resistance in HIV infected pregnant women. The effectiveness of short-term (7 day therapy) versus long-term (21-day therapy) regimens will also be compared.

The study hypotheses are: 1) intrapartum SD NVP with a 21-day course of antiretroviral therapy (ART) results in less frequent selection of NVP-resistant HIV-1 variants than intrapartum SD NVP with a 7-day course of ART, and 2) a 7- or 21-day course of lamivudine/zidovudine (3TC/ZDV), emtricitabine/tenofovir disoproxil fumarate (FTC/TDF), or lopinavir/ritonavir (LPV/r) following SD NVP will not select nucleoside reverse transcriptase inhibitor (NRTI)- or protease inhibitor (PI)- resistant HIV-1 variants.

DETAILED DESCRIPTION:
A major disadvantage of giving SD NVP is the potential for maternal development of NVP resistance and additional resistance to other nonnucleoside reverse transcriptase inhibitors (NNRTI) in the mother; as a result, future treatment options may be limited for these HIV infected women. The purpose of the study is to determine which of three ART regimens most effectively deters the development of maternal NVP resistance in HIV infected pregnant women postpartum. This study also compared the effectiveness of short-term versus long-term ART in discouraging the development of maternal NVP resistance.

Some mothers in this study received ZDV monotherapy prior to SD NVP administration; initiation of ZDV monotherapy was at the discretion of the site investigator and was be provided by this study. Randomization was stratified by receipt of ZDV monotherapy during the pregnancy.

Prior to labor, mothers were randomly assigned to receive SD NVP at the onset of labor and one of three postpartum ART regimens: 3TC/ZDV, FTC/TDF, and LPV/r. In addition, participants were randomly assigned to receive 7 or 21 days of their assigned postpartum treatment.

Mothers were followed for 96 weeks following delivery; there were 11 study visits for mothers during the study. At the onset of labor, medical and medication history, a targeted physical exam, and an obstetrical exam occurred. Additional physical exams occurred on Day 1 and Weeks 1 and 3. Blood collection occurred at 8 study visits between Weeks 3 and 96. Infants were followed for up to 96 weeks after birth; there were 8 study visits for infants during the study. Infants who had ever been breastfed had study visits at Weeks 16, 24, 48, and 96, and at about 1 and 2 years of age. A physical exam, medication history, and blood collection occurred at each infant visit. Mothers and infants could be prescribed continuing ART, but such ART was be provided by this study.

ELIGIBILITY:
Inclusion Criteria for Mothers:

* HIV-1 infected
* CD4 count 250 cells/mm3 or greater within 30 days of study entry
* The following laboratory values obtained within 30 days prior to study entry: absolute neutropil count >= 750/mm3; hemoglobin >= 8.0 g/dL; platelet count >= 50,000/mm3; calculated creatinine clearance (Cockcroft-Gault formula) > 60 mL/min; AST(SGOT) and ALT(SGPT) < 5 x ULN; total bilirubin < 1.5 X ULN.
* Pregnant with a viable fetus at 28 to 38 weeks gestation at study entry.
* Willing to give birth to baby in a hospital or clinic
* Written informed consent from parent or guardian, if applicable

Exclusion Criteria for Mothers:

* Any ART, including single-dose NVP, prior to study entry. Mothers who receive ZDV monotherapy prior to labor under the supervision of the site investigator are not excluded.
* Known allergy or sensitivity to study drugs or their formulations
* Current drug or alcohol abuse that may interfere with the study
* Serious illness requiring systemic treatment or hospitalization. Participants who complete therapy or are clinically stable on therapy for at least 14 days prior to study entry are not excluded.
* Hepatitis B surface antigen positive within 180 days prior to study entry
* Active tuberculosis infection requiring treatment
* Prior enrollment in this study
* Expect to use ART, except ZDV monotherapy, prior to onset of labor
* Expect to use ART other than study medications from delivery to 9 weeks postpartum

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2006-03; Primary Completion 2010-04 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Hitti, MD, MPH, Study Chair — Department of Obstetrics/Gynecology, Perinatal Medicine, University of Washington Medical Center; Deborah McMahon, MD, Study Chair — Division of Infectious Diseases, Department of Medicine, University of Pittsburgh
Locations (8):
- Les Centres GHESKIO Clinical Research Site (GHESKIO-INLR) CRS, Port-au-Prince, Haiti
- India (2):
  - Byramjee Jeejeebhoy Government Medical College CRS, Pune, Maharashtra
  - Chennai Antiviral Research and Treatment (CART) CRS, Chennai, Tamil Nadu
- Blantyre CRS, Blantyre, Malawi
- South Africa (2):
  - Wits Helen Joseph Hospital CRS (Wits HJH CRS), Johannesburg, Gauteng
  - Durban International CRS, Westville, KwaZulu-Natal
- Kilimanjaro Christian Medical CRS, Moshi, Tanzania
- Joint Clinical Research Center (JCRC)/Kampala CRS, Kampala, Uganda

REFERENCES:
- [Background] Cunningham CK, Chaix ML, Rekacewicz C, Britto P, Rouzioux C, Gelber RD, Dorenbaum A, Delfraissy JF, Bazin B, Mofenson L, Sullivan JL. Development of resistance mutations in women receiving standard antiretroviral therapy who received intrapartum nevirapine to prevent perinatal human immunodeficiency virus type 1 transmission: a substudy of pediatric AIDS clinical trials group protocol 316. J Infect Dis. 2002 Jul 15;186(2):181-8. doi: 10.1086/341300. Epub 2002 Jun 26. PMID 12134253
- [Background] Eshleman SH, Jackson JB. Nevirapine resistance after single dose prophylaxis. AIDS Rev. 2002 Apr-Jun;4(2):59-63. PMID 12152519
- [Background] Jourdain G, Ngo-Giang-Huong N, Le Coeur S, Bowonwatanuwong C, Kantipong P, Leechanachai P, Ariyadej S, Leenasirimakul P, Hammer S, Lallemant M; Perinatal HIV Prevention Trial Group. Intrapartum exposure to nevirapine and subsequent maternal responses to nevirapine-based antiretroviral therapy. N Engl J Med. 2004 Jul 15;351(3):229-40. doi: 10.1056/NEJMoa041305. Epub 2004 Jul 9. PMID 15247339
- [Background] Lyons FE, Coughlan S, Byrne CM, Hopkins SM, Hall WW, Mulcahy FM. Emergence of antiretroviral resistance in HIV-positive women receiving combination antiretroviral therapy in pregnancy. AIDS. 2005 Jan 3;19(1):63-7. doi: 10.1097/00002030-200501030-00007. PMID 15627034
- [Background] Sullivan JL. Prevention of mother-to-child transmission of HIV--what next? J Acquir Immune Defic Syndr. 2003 Sep;34 Suppl 1:S67-72. doi: 10.1097/00126334-200309011-00010. PMID 14562860
- [Result] McMahon D, Noel F, Zheng L, Kabanda J, Halvas E, Taulo F, Kumarasamy N, Wallis C, Hughes M, Mellors J. Suppression of NVP Resistance with 7- vs 21-day ARV Regimens after Single-dose NVP: Results of A5207. Presented at 18th Conference on Retroviruses & Opportunistic Infections (CROI 11) on 03/01/2011 at Boston, MA
- [Result] Hong F, Halvas E, Chan E, Zheng L, Hughes M, Hitti J, McMahon D, Mellors J. Suppression of Minor NVP-Resistant Variants With 7- vs. 21-Day Antiretroviral Regimens After Single Dose Nevirapine. Presented at 20th Anniversary of the International Workshop on HIV & Hepatitis Virus Drug Resistance and Curative Strategies on Jun 9, 2011, Los Cabos, Mexico
- [Derived] McMahon DK, Zheng L, Hitti J, Chan ES, Halvas EK, Hong F, Kabanda J, Taulo F, Kumarasamy N, Bonhomme J, Wallis CL, Klingman KL, Hughes MD, Mellors JW. Greater suppression of nevirapine resistance with 21- vs 7-day antiretroviral regimens after intrapartum single-dose nevirapine for prevention of mother-to-child transmission of HIV. Clin Infect Dis. 2013 Apr;56(7):1044-51. doi: 10.1093/cid/cis1219. Epub 2013 Jan 8. PMID 23300238

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited at 8 sites: 2 from South Africa, 2 from India, and 1 each from Haiti, Uganda, Tanzania, and Malawi, between January 2007 to October 2009.
Pre-assignment Details: 62 participants who randomized but did not start study treatment were excluded from the analysis. These 62 participants were either off study prior to delivery or delivered on study but did not take any dose of study treatment.
  All the analyses were restricted to the 422 women who received study treatment.
Groups:
- 7-day Lamivudine/Zidovudine (3TC/ZDV): SD NVP and 3TC/ZDV provided at onset of active labor, followed by 7 days of 3TC/ZDV.
- 21-day Lamivudine/Zidovudine (3TC/ZDV): SD NVP and 3TC/ZDV provided at onset of active labor, followed by 21 days of 3TC/ZDV.
- 7-day Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF): SD NVP and FTC/TDF provided at onset of active labor, followed by 7 days of FTC/TDF.
- 21-day Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF): SD NVP and FTC/TDF provided at onset of active labor, followed by 21 days of FTC/TDF.
- 7-day Lopinavir/Ritonavir (LPV/r); 21-day Lopinavir/Ritonavir (LPV/r): SD NVP and LPV/r provided at onset of active labor, followed by 7 days of LPV/r.
Period: Overall Study
Arm/Group | 7-day Lamivudine/Zidovudine (3TC/ZDV) | 21-day Lamivudine/Zidovudine (3TC/ZDV) | 7-day Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) | 21-day Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) | 7-day Lopinavir/Ritonavir (LPV/r) | 21-day Lopinavir/Ritonavir (LPV/r)
Started | 73 | 68 | 75 | 67 | 71 | 68
Completed | 72 | 67 | 72 | 66 | 70 | 66
Not Completed | 1 | 1 | 3 | 1 | 1 | 2
Not completed — Lost to Follow-up | 1 | 0 | 3 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 7-day Lamivudine/Zidovudine (3TC/ZDV) | 21-day Lamivudine/Zidovudine (3TC/ZDV) | 7-day Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) | 21-day Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) | 7-day Lopinavir/Ritonavir (LPV/r) | 21-day Lopinavir/Ritonavir (LPV/r) | Total
Number analyzed (Participants) | 73 | 68 | 75 | 67 | 71 | 68 | 422
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (6) | 27 (5) | 26 (5) | 26 (5) | 27 (6) | 26 (5) | 27 (5)
Age, Customized [Number; unit: participants]
  Between 13 and 19 years | 2 | 1 | 5 | 3 | 3 | 3 | 17
  Between 20 and 29 years | 49 | 46 | 53 | 46 | 47 | 48 | 289
  Between 30 and 39 years | 20 | 20 | 16 | 18 | 19 | 16 | 109
  >= 40 years | 2 | 1 | 1 | 0 | 2 | 1 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 68 | 75 | 67 | 71 | 68 | 422
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Haiti | 12 | 11 | 10 | 7 | 9 | 9 | 58
  Tanzania | 3 | 1 | 3 | 3 | 2 | 2 | 14
  Uganda | 17 | 16 | 18 | 17 | 17 | 16 | 101
  South Africa | 13 | 8 | 10 | 9 | 10 | 10 | 60
  Malawi | 13 | 14 | 14 | 12 | 17 | 15 | 85
  India | 15 | 18 | 20 | 19 | 16 | 16 | 104
Gestational age at NVP dosing, Continuous [Mean (Standard Deviation); unit: weeks] | 38 (2) | 39 (2) | 38 (2) | 38 (3) | 38 (2) | 38 (2) | 38 (2)
Screening CD4 count Categorical [Number; unit: participants]
  250-349 cells/mm^3 | 15 | 7 | 8 | 6 | 20 | 13 | 69
  350-499 cells/mm^3 | 24 | 21 | 29 | 29 | 25 | 22 | 150
  >=500 cells/mm^3 | 34 | 40 | 38 | 32 | 26 | 33 | 203
Screening CD4 count Continuous [Mean (Standard Deviation); unit: cells/mm^3] | 538 (244) | 585 (215) | 537 (186) | 545 (191) | 505 (205) | 566 (249) | 545 (216)
Screening HIV-1 RNA Categorical [Number; unit: participants]
  <=400 copies/mL | 17 | 13 | 13 | 12 | 12 | 16 | 83
  401-999 copies/mL | 12 | 8 | 7 | 11 | 6 | 4 | 48
  1000-9999 copies/mL | 17 | 26 | 33 | 25 | 29 | 18 | 148
  10000-99999 copies/mL | 17 | 17 | 18 | 14 | 20 | 26 | 112
  100000-749999 copies/mL | 8 | 3 | 4 | 5 | 4 | 4 | 28
  >=750000 copies/mL | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Missing/Unknown | 1 | 1 | 0 | 0 | 0 | 0 | 2
Screening HIV-1 RNA Continuous [Mean (Standard Deviation); unit: log10 copies/mL] | 3.50 (1.01) | 3.55 (0.90) | 3.54 (0.82) | 3.50 (0.88) | 3.63 (0.90) | 3.66 (0.92) | 3.56 (0.90)
Actual ZDV exposure during pregnancy [Number; unit: participants]
  yes | 46 | 47 | 47 | 42 | 43 | 42 | 267
  no | 27 | 21 | 28 | 25 | 28 | 26 | 155

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With New Circulating Nonnucleoside Reverse Transcriptase Inhibitor (NNRTI)-Resistant Variants as Detected by Standard Composite (Bulk) Genotyping
Description: For the 7-day treatment duration group, only the genotype results from weeks 3 and 7 contributed to the primary endpoint; For the 21-day treatment duration groups, only the genotype results from weeks 5 and 9 contributed to primary endpoint.
  10 participants who did not have resistance samples available were excluded from the primary endpoint analysis.
Time Frame: 2 and 6 weeks after completion of treatment
Population: 412 women with primary endpoint results available
Measure: Number; unit: participants
Arm/Group | 7-day Lamivudine/Zidovudine (3TC/ZDV) | 21-day Lamivudine/Zidovudine (3TC/ZDV) | 7-day Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) | 21-day Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) | 7-day Lopinavir/Ritonavir (LPV/r) | 21-day Lopinavir/Ritonavir (LPV/r)
Number analyzed (Participants) | 73 | 67 | 71 | 65 | 71 | 65
participants | 1 | 0 | 0 | 0 | 3 | 1
Statistical Analysis 1: Comparison: 7-day Lamivudine/Zidovudine (3TC/ZDV) vs 21-day Lamivudine/Zidovudine (3TC/ZDV) vs 7-day Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) vs 21-day Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) vs 7-day Lopinavir/Ritonavir (LPV/r) vs 21-day Lopinavir/Ritonavir (LPV/r); Compare proportion of women with new NNRTI-resistant variants between treatment durations (7-day vs. 21 day), pooled over ARV regimens (3TC/ZDV, FTC/TDF, and LPV/r), stratified by ARV regimen and the actual receipt of antenatal ZDV; Test type: Superiority or Other; p = 0.37, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by ARV regimen and the actual receipt of antenatal ZDV
Statistical Analysis 2: Comparison: 7-day Lamivudine/Zidovudine (3TC/ZDV) vs 21-day Lamivudine/Zidovudine (3TC/ZDV) vs 7-day Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) vs 21-day Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) vs 7-day Lopinavir/Ritonavir (LPV/r) vs 21-day Lopinavir/Ritonavir (LPV/r); Compare proportion of women with new NNRTI-resistant variants among ARV regimens (3TC/ZDV vs. FTC/TDF vs. LPV/r), pooled over treatment durations 7-day and 21-day, stratified by treatment duration and the actual receipt of antenatal ZDV; Test type: Superiority or Other; p = 0.091, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by treatment duration and the actual receipt of antenatal ZDV

2. Secondary Outcome: Number of Participants With New Circulating NRTI-resistant Variants Detected by Standard Composite (Bulk) Genotyping.
Description: For the 7-day treatment duration group, only the genotype results from weeks 3 and 7 contributed; For the 21-day treatment duration groups, only the genotype results from weeks 5 and 9 contributed.
Time Frame: 2 and 6 weeks after completion of treatment
Measure: Number; unit: participants
Arm/Group | 7-day Lamivudine/Zidovudine (3TC/ZDV) | 21-day Lamivudine/Zidovudine (3TC/ZDV) | 7-day Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) | 21-day Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) | 7-day Lopinavir/Ritonavir (LPV/r) | 21-day Lopinavir/Ritonavir (LPV/r)
Number analyzed (Participants) | 73 | 67 | 71 | 65 | 71 | 65
participants | 0 | 1 | 1 | 1 | 1 | 0

3. Secondary Outcome: Number of Participants With New PI-resistant Variants as Detected by Standard Composite (Bulk) Genotyping.
Description: as for outcome 2
Time Frame: 2 and 6 weeks after completion of treatment
Measure: Number; unit: participants
Arm/Group | 7-day Lamivudine/Zidovudine (3TC/ZDV) | 21-day Lamivudine/Zidovudine (3TC/ZDV) | 7-day Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) | 21-day Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) | 7-day Lopinavir/Ritonavir (LPV/r) | 21-day Lopinavir/Ritonavir (LPV/r)
Number analyzed (Participants) | 73 | 67 | 71 | 65 | 71 | 65
participants | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Severe (Grade 3) and Higher Adverse Events and Any Grade Adverse Event That Leads to a Treatment Change From First Day of Study Treatment to Week 12
Description: Grade 3 or higher signs and symptoms, laboratory abnormalities, events that are reported through the EAE system, and any grade event that leads to a treatment change from first day of study treatment to week 12.
  Grade 3 = Severe Grade 4 = Life threatening Grade 5 = Death
Time Frame: From first day of study treatment to week 12
Measure: Number; unit: participants
Arm/Group | 7-day Lamivudine/Zidovudine (3TC/ZDV) | 21-day Lamivudine/Zidovudine (3TC/ZDV) | 7-day Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) | 21-day Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) | 7-day Lopinavir/Ritonavir (LPV/r) | 21-day Lopinavir/Ritonavir (LPV/r)
Number analyzed (Participants) | 73 | 68 | 75 | 67 | 71 | 68
participants | 5 | 1 | 1 | 0 | 2 | 2

5. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Prematurely
Description: participants assigned to 7-day treatment arm and 21-day treatment arm were supposed to stay in study treatment for 7 days and 21 days respectively.
Time Frame: From first day of study treatment to last day of study treatment (up to 21 days)
Measure: Number; unit: participants
Arm/Group | 7-day Lamivudine/Zidovudine (3TC/ZDV) | 21-day Lamivudine/Zidovudine (3TC/ZDV) | 7-day Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) | 21-day Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) | 7-day Lopinavir/Ritonavir (LPV/r) | 21-day Lopinavir/Ritonavir (LPV/r)
Number analyzed (Participants) | 73 | 68 | 75 | 67 | 71 | 63
participants | 0 | 2 | 0 | 0 | 0 | 5

ADVERSE EVENTS:
Time Frame: From first treatment date to 12 weeks of follow up.
Description: Expedited adverse event(AE) reporting followed intensive DAIDS Reporting Level, which included AEs resulting in death, congenital anomalies, fetal losses, significant disabilities, requiring hospitalization, and >=3 grade 3 AEs defined by the "DAIDS Table for Grading the Severity of Adult and Pediatric AEs".
Groups:
- 21-day LPV/r: SD NVP and LPV/r provided at onset of active labor, followed by 21 days of LPV/r
Arm/Group | 7-day 3TC/ZDV | 21-day 3TC/ZDV | 7-day FTC/TDF | 21-day FTC/TDF | 7-day LPV/r | 21-day LPV/r
Serious Adverse Events (participants affected / at risk) | 2/73 | 0/68 | 1/75 | 0/67 | 1/71 | 0/68
Other Adverse Events (participants affected / at risk) | 0/73 | 0/68 | 0/75 | 0/67 | 0/71 | 0/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 7-day 3TC/ZDV (N=73) | 21-day 3TC/ZDV (N=68) | 7-day FTC/TDF (N=75) | 21-day FTC/TDF (N=67) | 7-day LPV/r (N=71) | 21-day LPV/r (N=68)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Uterine rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 1 | 0
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights